CLINICAL TRIAL: NCT00698724
Title: A Prospective, Randomized Single-Masked Clinical Trial Comparing OCT and Visual Acuity Outcomes in Subjects Undergoing Cataract Surgery, Who Receive Xibrom Ophthalmic Solution and Standard Presurgical Care vs. Xibrom Ophthalmic Solution Plus Prednisolone Acetate 1% and Standard Presurgical Care
Brief Title: Comparing Optical Coherence Tomography (OCT) and Visual Acuity Outcomes in Subjects Undergoing Cataract Surgery, Who Receive Xibrom Ophthalmic Solution and Standard Presurgical Care vs. Xibrom Ophthalmic Solution Plus Prednisolone Acetate 1% and Standard Presurgical Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bp Consulting, Inc (Network)
Responsible Party: Dr. Gills, St. Luke's Cataract and Laser Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5359
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2009-06-10 (Estimated); Status verified 2009-06

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract | interventions — bromfenac; prednisolone acetate

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Active Comparator): Group 1: Xibrom, Optive
  Interventions: Drug: Xibrom, and Optive
- 2 (Active Comparator): Group 2: Xibrom, Pred Forte
  Interventions: Drug: Xibrom and Pred Forte

INTERVENTIONS:
Drug: Xibrom, and Optive — Xibrom: two drops a day, three days before surgery and 21 days after surgery. Optive: three times a day for 21 days after surgery.
  Arms: 1
Drug: Xibrom and Pred Forte — Xibrom: two drops a day, three days before surgery and 21 days after surgery. Pred Forte: three times a day for 21 days after surgery.
  Arms: 2

SUMMARY:
To compare the efficacy of twice-daily topical bromfenac (Xibrom) ophthalmic solution alone versus twice-daily topical Xibrom with prednisolone acetate 1% three-times daily on visual acuity and OCT measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age.

  * Expectation of 20/25 best corrected visual acuity (BCVA) post-operatively.
  * Patients should be in good general health and devoid of recognized risk factors for CME.
  * Patients with systemic diseases are eligible only if there were no ocular manifestations of the disease (specifically diabetics without retinopathy)
  * Patients must be likely to provide informed consent, take study medications as directed, and complete all study visits
  * Only one eye of each treated patient may be included in the study

Exclusion Criteria:

* Any known contraindications to any study medication or their component
* Presence of uncontrolled systemic disease
* Required use of other ocular medications during the study

  o Artificial tears may be used
* Diabetics with any clinically evident or history of retinopathy
* Individuals with age-related macular changes, epi-retinal membranes, other retino-vascular diseases and/or other macular disorders thought to have a less than 20/25 surgical outcome expectation
* Abnormal pre-operative OCT (if obtainable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
OCT | 2-4 months

SECONDARY OUTCOMES:
Visual Acuity | 2-4 months

CONTACTS AND LOCATIONS:
Overall Officials: James Gills, MD, Principal Investigator — St. Luke's Cataract and Laser Institute
Locations (1):
- St. Luke's Cataract and Laser institute, Tarpon Springs, Florida, United States